CLINICAL TRIAL: NCT07363837
Title: A Randomized, Double-blind, Placebo/Positive Control, Dose-finding Phase Ib/IIa Clinical Trial Evaluating the Safety, Tolerability, and Pharmacokinetics of SIBP-A16 Injection in Premature Infants and Full-term Infants
Brief Title: Phase Ib/IIa Clinical Trial of SIBP-A16 Injection in Premature Infants and Full-term Infants
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-A16-002
Record Dates: First submitted 2026-01-05; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: RSV; Preliminary efficacy; Premature and term infants; Pharmacokinetics; Safety; Tolerability
MeSH Terms: conditions — Premature Birth | interventions — nirsevimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): SIBP-A16 injection
  Interventions: Drug: SIBP-A16 injection
- Positive Comparator (Active Comparator): Nirsevimab
  Interventions: Drug: Nirsevimab
- Placebo (Placebo Comparator): SIBP-A16 buffer solution
  Interventions: Drug: SIBP-A16 buffer solution

INTERVENTIONS:
Drug: SIBP-A16 injection — Strength: dose 1, dose 2 and dose 3. Single administration via intramuscular or intravenous injection.
  Arms: Experimental group
Drug: Nirsevimab — Participants will receive one dose of Nisibimab via intramuscular injection.
  Arms: Positive Comparator
Drug: SIBP-A16 buffer solution — Participants in the placebo group will be assigned to four dose cohorts, and they will receive one dose of Placebo via intramuscular injection.
  Arms: Placebo

SUMMARY:
This trial employs a randomized, double-blind, placebo/positive control, and dose-finding design to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of SIBP-A16 injection in premature and term infants.

DETAILED DESCRIPTION:
This study established three study groups: the test drug group, the placebo group, and the positive control group. Four dose cohorts were set up: Cohort 1 (Dose 1), Cohort 2 (Dose 2), Cohort 3 (Dose 3), and Cohort 4 (Dose 2). A total of 36 participants were enrolled. The drug will be administered via intramuscular injection as a single dose. Initially, Cohort 1 enrolled 7 participants, who were randomly assigned to receive either one dose of the test drug or placebo. After completing the initial 14-day safety observation, if the dose escalation termination criteria were not triggered, participants were enrolled into Cohort 2 (11 participants, randomly assigned to receive either one dose of the test drug or placebo). Once Cohort 2 was fully enrolled, participants could be enrolled into Cohort 4 (7 participants, randomly assigned to receive either one dose of the positive control drug or placebo). After Cohort 2 completed the 14-day safety observation, participants were enrolled into Cohort 3 (11 participants, randomly assigned to receive either one dose of the test drug or placebo) following the same procedure. If the dose escalation termination criteria were triggered, the Data Monitoring Committee (DMC) would conduct a safety assessment and discuss with the research team and sponsor whether to terminate the dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* During screening, infants within 1 year of age, including premature infants (gestational age ≥29 to <35 weeks) and full-term infants (gestational age ≥35 weeks), with underlying diseases but no other risk factors, are allowed to participate in the trial;
* Infants with a body weight ≥3 kg at screening;
* Infants who are entering their first RSV infection season at screening;
* Parents/legal guardians of trial participants have signed the informed consent form;
* Parents/legal guardians of trial participants are able to understand and comply with the requirements and procedures of the protocol, including scheduled center visits, telephone interviews, and blood sample collection;
* Participants can complete the follow-up period, which is approximately 1 year after the administration of the study drug.

Exclusion Criteria:

* Any fever (≥37.5°C, axillary temperature) or acute illness (defined as the presence of moderate or severe symptoms or signs) occurring within 7 days prior to drug administration;
* Having experienced Lower Respiratory Tract Infections (LRTI) within the previous 7 days prior to randomization, or having active LRTI at the time of randomization;
* Individuals with chronic eczema or urticaria, or those with an allergic constitution who are allergic to multiple drugs, or those with a known history of allergy to immunoglobulin products, blood products, other exogenous proteins, or any components of this product;
* Had a history of RSV infection before randomization, or had active RSV infection at the time of randomization;
* Those who have received non-oral inactivated vaccines or component vaccines within 7 days before administration;
* Having received a non-oral live attenuated vaccine within 30 days prior to drug administration;
* Participants who have received any medication within 7 days prior to drug administration, except for: a) various vitamins and iron supplements; b) systemic over-the-counter medications (such as analgesics) for common pediatric symptoms, which may be used occasionally, as determined by the investigator;
* Participants with autoimmune diseases who are currently receiving, or are expected to receive according to the investigator's judgment, immunosuppressive therapy (including steroids, excluding topical steroids) during the trial period;
* Have previously used or are expected to receive blood products or immunoglobulin products during the trial period;
* Known renal dysfunction or liver dysfunction;
* Known to have chronic lung disease (CLD)/bronchopulmonary dysplasia;
* Congenital respiratory abnormalities with clinical significance;
* Suffering from congenital heart disease (CHD) accompanied by significant hemodynamic changes;
* Suffering from chronic epilepsy or progressive or unstable neurological disorders;
* Those who have previously experienced or are suspected to have experienced life-threatening acute events, and are still deemed unsuitable for participating in clinical trials by the researchers;
* Known immune deficiency, including infection with human immunodeficiency virus (HIV);
* The mother is infected with HIV (unless it has been proven that the trial participant is not infected);
* The mother received the RSV vaccine during pregnancy;
* Have received any investigational drugs or participated in any intervention studies;
* Any other circumstances that the researcher believes may interfere with the evaluation of the study drug or the interpretation of the study results;
* The participants are the children of the researchers, their subordinate researchers, relatives, or staff members of the sponsor.

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
AE (Adverse Events) | From day 1 to day 360 after administration
  That is adverse events, any adverse events that occurred to the participant during the study period.
SAE (Serious Adverse Events) | From day 1 to day 360 after administration
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.
Adverse Event of Special Interest (AESI) | From day 1 to day 360 after administration
  Adverse events defined in the protocol that require special attention, such as abnormal liver function, anaphylactic reaction, hypersensitivity reaction, etc.
New-onset chronic diseases (NOCD) | From day 1 to day 360 after administration
  NOCD refer to chronic non-communicable diseases that emerge during clinical trials.

SECONDARY OUTCOMES:
AUC (Area Under The Plasma Concentration Versus Time Curve) | Before injection, on the 7th, 30th, 90th, 150th and 360th days after administration
  It shows the degree to which a drug is absorbed and used in the body.
Cmax (Peak Plasma Concentration) | Before injection, on the 7th, 30th, 90th, 150th and 360th days after administration
  It shows the highest plasma concentration of a drug that can be achieved after administration.
Tmax (Peak Time) | Before injection, on the 7th, 30th, 90th, 150th and 360th days after administration
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the participant plasma concentration curve after administration.
Detecting RSV neutralizing antibody activity at various time points | Before injection, on the 7th, 30th, 90th, 150th and 360th days after administration
  The RSV neutralizing assay was used to analyze the neutralizing activity of participants against RSV at various time points (before administration, and on days 7, 30, 90, 150, and 360 after administration).
Level of Anti-drug antibody (ADA) | Before injection, on the 30th, 150th and 360th days after administration
  If ADA is positive, further use validated analytical methods to detect the anti-SIBP-A16 neutralizing antibody (Nab).

CONTACTS AND LOCATIONS:
Overall Officials: Hanwen Liu, Principal Investigator — West China Second Hospital, Sichuan University
Locations (1):
- West China Second Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No